CLINICAL TRIAL: NCT05129982
Title: Reliability of Methods for Determining the Vibration Threshold That Triggers the Reflex
Brief Title: Reliability of Methods for Determining the Vibration Threshold
Acronym: IPMTRH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: WBVsensor
Record Dates: First submitted 2021-11-08; First posted 2021-11-22 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Reflex, Abnormal
Keywords: sensor; vibration; reflex
MeSH Terms: conditions — Reflex, Abnormal

STUDY DESIGN:
Intervention Model Description: self-controlled study
Masking Description: With the cumulative average method, latency estimation will be made blindly.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): The reflex response will be recorded during whole-body vibration.
  Interventions: Device: whole body vibration

INTERVENTIONS:
Device: whole body vibration — whole body vibration is a modality of physical therapy

SUMMARY:
It is known that whole-body vibration (TVV) has beneficial neuromuscular effects such as muscle strength increase. These beneficial effects are explained by the muscular reflex response induced by TVV. Reflex latency measurement is frequently used in clinical and neurophysiological research. The latency of the reflex response induced by TVV is defined as the period between the onset of the vibration stimulus and the onset point of the spike in the EMG signal. The current research aimed to determine whether the cumulative average method is reliable for estimating the EST.

DETAILED DESCRIPTION:
This is an experimental study for method development; a self-controlled (single group) study. Ten healthy male or female subjects between the ages of 18-45 will be included in the study. After obtaining informed consent from the subjects, 30 Hz low amplitude (2 mm) vibration for 30 seconds will be applied on the PowerPlate Pro5 device to meet TVV. After three minutes of rest, two sets of TVV will be applied for test purposes. For the test TVV, vibration will be applied at 25, 30, 35, 40, 45, 50 Hz frequencies, each lasting 30 seconds, with low amplitude.

Vibration stimuli detected by using an accelerometer fixed on the TVV platform will be recorded the Data acquisition (PowerLab data acquisition system (ADInstruments, Oxford, United Kingdom). Soleus EMG responses will be recorded using the superficial electrodes (Kendall Covidien). The sample rate for recordings will be 40KHz.

Latency calculation with Cumulative Average Method: It will be done. An 80-500 Hz band-pass filter and full-wave rectification will be applied to EMG recordings. The peak of reflex responses (spike) will be marked with the help of LabChart7 (ver 7.3.7, ADInstruments, Oxford, United Kingdom). According to this marked point, the averaging process covered 75 ms of the vibration data preceding the trigger and 15 ms after for each vibration frequency separately. Then, the average of the five vibration frequencies will be calculated for the accelerometer recordings and EMG recordings. The point where the standard error is lowest in the accelerometer recordings will be determined as the "effective stimulation point".

ELIGIBILITY:
Inclusion Criteria:

* Both gender
* 20-40 aged
* Healthy volunteer

Exclusion Criteria:

* People with any health problems

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2021-12-13 (Actual)

PRIMARY OUTCOMES:
Threshold vibration stimulus | A single point in time (1 day)
  Threshold vibration stimulus intensity that activates the reflex response

CONTACTS AND LOCATIONS:
Overall Officials: İLHAN KARACAN, Principal Investigator — Istanbul Physical Medicine Rehabilitation Training & Research Hospital
Locations (1):
- Istanbul Physical Medicine Rehabilitation Training & Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are available from the corresponding author upon reasonable request.